CLINICAL TRIAL: NCT01699698
Title: Pancreatic Juice Diagnosis From Duodenum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olympus Corporation (Industry)
Collaborators: Mayo Clinic (Other); Kyushu University (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: OMSC-PJD-1
Record Dates: First submitted 2012-09-24; First posted 2012-10-04 (Estimated); Results first posted 2015-09-03 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic adenocarcinoma
MeSH Terms: interventions — Biomarkers, Tumor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Test subject (Experimental)
  Interventions: Other: Tumor markers

INTERVENTIONS:
Other: Tumor markers — Duodenal juice are collected using endoscope and cannula. Tumor markers of collected samples are analyzed. The marker concentration is applied to statistical analysis.

SUMMARY:
Purpose of this study is to understand the clinical feasibility of duodenal juice diagnosis to screen UICC stage II pancreatic ductal adenocarcinoma patients.

DETAILED DESCRIPTION:
Pancreatic cancer (PC) is the most lethal of all major cancers with a five year survival rate of 5 %. While stage I and II tumors leads to an improvement in survival, almost all PCs are currently diagnosed at more advanced non-resectable stages since minimally invasive technique which is capable of screening early-stage PC does not exist. Serum CA19-9 is not recommended as a screening technique because of its low sensitivity and specificity. Imaging modalities such as MRI, CT, EUS and ERCP are more accurate but are not appropriate screening tools due to their high cost, discomfort and complications. Therefore, there is a strong demand for a screening tool with high sensitivity and specificity which is highly acceptable for the patient.

The investigators would like to standardize the detection method of pancreatic cancer that uses the duodenal juice as an optional endoscopic diagnosis. It's a very useful chance to collect pancreatic juice from duodenum, it is called "duodenal juice" ,if we collect them without additional invasion. The investigators would like to collect duodenal juice during undergoing upper gastrointestinal endoscopy and analyze the pancreatic tumor markers in duodenal juice. A definite diagnosis of the patient is made with histology, cytology or imaging diagnosis and the result of each definite diagnosis is correlated to the each marker analyzing result of duodenal juice. Therefore this study can be positioned as a feasibility study to confirm clinical performance.

ELIGIBILITY:
Inclusion Criteria:

* Common inclusion criterion
* Age is 18 years or older.
* Informed consent was obtained.
* Inclusion criterion for normal cohort
* An upper GI endoscopy is scheduled to check upper abdominal symptoms.
* No findings of pancreatic disorder as documented by CT or MRI or EUS
* Inclusion criterion for PC suspicious cohort
* A EUS or ERCP is scheduled to suspected pancreatic disorder.

Exclusion Criteria:

* Common exclusion criterion
* Severe cardiac disease
* Severe respiratory disease
* Bleeding disorders
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Raimondo, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- Mayo Clinic Jacksonville, Jacksonville, Florida, United States
- Kyushu University, Fukuoka, Fukuoka, Japan

REFERENCES:
- [Background] Pungpapong S, Noh KW, Woodward TA, Wallace MB, Al-Haddad M, Raimondo M. Endoscopic ultrasound and IL-8 in pancreatic juice to diagnose chronic pancreatitis. Pancreatology. 2007;7(5-6):491-6. doi: 10.1159/000108966. Epub 2007 Oct 1. PMID 17912013

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Subject: UICC StageII pancreatic ductal adenocarcinoma cohort
- Control: Normal cohort
Period: Overall Study
Arm/Group | Test Subject | Control
Started | 44 | 61
Completed | 42 | 56
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Test Subject: UICC Stage II pancreatic ductal adenocarcinoma cohort
- Total: Total of all reporting groups
Arm/Group | Test Subject | Control | Total
Number analyzed (Participants) | 42 | 56 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 36 | 49
  >=65 years | 29 | 20 | 49
Age, Continuous [Median (Full Range); unit: years] | 70 [49 to 88] | 60 [23 to 81] | 64 [23 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 36 | 49
  Male | 29 | 20 | 49
Region of Enrollment [Number; unit: participants]
  United States | 20 | 28 | 48
  Japan | 22 | 28 | 50

OUTCOME MEASURES:

1. Primary Outcome: The Concentration of the Pancreatic Cancer Markers of the Normal Cohort and UICC Stage II Pancreatic Ductal Adenocarcinoma Cohort
Description: We hypothesized that there is a statistically-significant difference between two cohorts.
  The cancer marker is S100P.
Time Frame: 1year
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Test Subject | Control
Number analyzed (Participants) | 42 | 56
pg/ml | 99097 [7386 to 1985933] | 34095 [611 to 497630]
Statistical Analysis 1: Comparison: Test Subject vs Control; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: The Sensitivity and Specificity to Detect UICC Stage II Pancreatic Ductal Adenocarcinoma Among All Participants.
Description: Based on each analyzing result of pancreatic cancer markers and corresponding final diagnosis, a receiver operating characteristic (ROC) is evaluated. A cut-off is then chosen from this ROC curve to maximize both sensitivity and specificity.<Method>1. create an ROC curve using the measured concentrations, 2. set a threshold, 3. report how many patients in each group would are exceeded the threshold. (The rate of exceeded threshold in Test subject group is sensitivity, The rate of 1-(the rate of exceeded threshold in Control group) is specificity.)
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Test Subject | Control
Number analyzed (Participants) | 42 | 56
participants | 31 | 17

ADVERSE EVENTS:
Groups:
- Normal: Normal cohort
Arm/Group | Test Subject | Normal
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/56
Other Adverse Events (participants affected / at risk) | 0/42 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can ask PI to consider that PI delete Sponsor's confidential information from any publication or extend the publication for a certain time to seek patent protection, provided, however that, PI can publish or registry any other information in accordance with FDAAA.